CLINICAL TRIAL: NCT03510195
Title: The Effectiveness of the Medicorp House Officer (HO) Preparatory Course for Medical Graduates on Confidence, Readiness, and Psychological Well-Being: A Quasi-Experimental Study
Brief Title: Effectiveness of Medicorp HO Preparatory Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Aneesa Abdul Rashid, Principal Investigator, Universiti Putra Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: upm/uctc/900/3/2/ktgs0518012
Record Dates: First submitted 2018-04-08; First posted 2018-04-27 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Psychological Stress; Depressive Symptoms; Anxiety State; Motivation
MeSH Terms: conditions — Stress, Psychological; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEDICORP HO PREPARATORY MODULE (Experimental): The participants that will have intervention which is the module
  Interventions: Other: MEDICORP HO PREPARATORY MODULE

INTERVENTIONS:
Other: MEDICORP HO PREPARATORY MODULE — 3 DAY course module to prepare medical graduates to become house officers

SUMMARY:
After completion of 5 years of medical school training, the next step of becoming a House Officer is said to be associated with high levels of stress. It has been associated with mental health problems amongst HOs and sometimes quitting the medical line altogether. In Malaysia, the number of HOs not completing housemanship training within the allocated time is slowly declining from 86.4% (2009) to 58.8% (2012). The dropout rate is said to be increasing yearly.

This causes a lot of constraints on the HO, their family, sponsors, patients and also the country. Amongst the reason for stress is the feeling of incompetency or "fear of making mistakes". Other work-related issues include workload, time management, financial, colleague and superior related issues.

Medicorp is a company that specializes in training for junior doctors and has come up with a module to help medical graduates cope with these issues. The module is a 3-day-course named the HO Preparatory Course. It was initially the brainchild of the Islamic Medical Association of Malaysia (IMAM) but was later privatized to accommodate the demand and the running of the module and courses. The module has been re-evaluated through feedback of participants and trainers to cater to the needs and wants of the newly graduate; be it local or overseas.

Therefore, the investigators would like to assess whether this intervention module is effective in addressing HO stress, therefore consequently reduce the risk of drop out and extension in HO training.

DETAILED DESCRIPTION:
METHODOLOGY

Study Setting:

This study will be conducted in International Youth Centre, Cheras. It has been the main focal point of where most of the courses have been conducted. It is within easy reach and centrally located near National University of Malaysia Hospital. Many participants will come from all around Malaysia to attend. The centre is equipped with a lecture hall and boarding for the participants.

Study Design:

This is a pre-post quasi-experimental study that will be conducted over 12 months duration. Participants in this study will undergo a House Officer (HO) preparatory course. The level of confidence, readiness and psychological wellbeing will be evaluated. There will be three assessment time points: at baseline (before the course), immediately after the course (only for level of confidence and readiness) and 1 month after working as HO. This study is unable to have a control because of constraints in resources.

Study Duration:

This study will start from April 2018 - March 2019

Sampling of participants:

Recruitment

Participants who attend the Medicorp HO Preparatory Course from April 2018 -March 2019 will be recruited into this study as the sampling frame. The eligibility criteria are based on the following:

The sampling methods employed in this study will be taking all participants who fulfill the eligibility criteria and agree to participate in this study.

Intervention:

The intervention in this study will be the Medicorp HO preparatory course which comprises of a 3-day training touching on aspects of HO training that is needed practically for an HO to function. The training will touch on the nature of the HO job, explaining about technical details such as the shift and on-call system. The tagging period, and assessments that HOs need to undergo during their training. They will be guided on how to clerk, review and present common as well as emergency cases. Other aspects involved in clerking such as common forms used in the wards and also how to refer cases is also discussed. Apart from that, soft skills such as communication among staff, financed, balancing social life and future career planning is incorporated in the training. There are hands-on training for participants for common procedures such as continuous bladder drainage insertion and venepuncture. The trainers are specialists, specialists in training, medical officers, and also house officers who come to share their experience. Medicorp encourages their alumni to be part of their training program. This module will be held on a 1-2 monthly basis. The Module Content is moderated by Medicorp based on discussions with the board of directors, advisors and feedback from participants. The training program is done as a lecture, tutorial and hands-on session. Before commencing the course, participants will be included in a WhatsApp group, for easier content sharing and updates of the course. They will continue this networking even after completion of this course. They will be also be guided in the online applications of their job through this application and also through Facebook. During the commencement of their job, Medicorp will use their database to guide them into different WhatsApp groups according to their place of work for additional support.

Sample size The sample size was calculated using G*Power 3.1 sample size calculator software. Based on reports by confidence score from a study analysing pre and post-emergency department posting in junior doctors was used. The mean overall confidence score was 56.475(24.67) at the end of month 1 and 62.775(28.69) at the end of month 4(Williams et al., 1997). The estimated sample size was 208 participants after accounting for the power of 80%, significance level of 0.05% and 30% attrition.

INSTRUMENTS AND DATA COLLECTION

Intervention: The Medicorp HO Preparatory Module

Tools for assessment:

1. Baseline questionnaire The study instrument will be a set of questionnaire that will be divided into sections A-E.

   The English versions will be used.
   1. Socio-demographic data :

      This will include certain details of participants such as:
      * Age
      * Sex
      * Religion
      * Ethnicity
      * Year of graduation
      * University of Graduation
      * Marital status
      * Place of work (evaluation during 1 month post HO-ship)
   2. Clinical Experience:

      This will be adapted from the International Medical University (IMU)Student Competency Survey. This will show participants past clinical experience on common procedures during their undergraduate years.
   3. Confidence level: Adapted from the IMU student competency questionnaire as explained in study outcome measures
   4. Readiness : Adapted from the IMU student competency questionnaire as explained in study outcome measures
   5. Psychological well -being : DASS as explained in study outcome measures
2. Post course questionnaire (immediate)

   1. Level of confidence
   2. Readiness
3. Case report form Conducted via telephone call at 1 month after starting work as HO Content will include

   1. Level of confidence
   2. Readiness
   3. DASS
   4. Work place information: which hospital and posting
   5. Any suggestions to improve the course based on your current working experience?

All the questionnaires will be pilot tested by testing this on 30 medical graduates before using the questionnaire.

Data collection

A pre-tested self-administered questionnaire which includes baseline socio-demography, adaptation of the IMU Student Competency Survey, and the Depression Anxiety Stress Scale will be used. 1 month follow-up will be done by telephone. After the participants have completed the course, their level of readiness and confidence will again be assessed via a self-administered questionnaire. This will be done on the last day of the course.

The participants will later be followed up 1 month after they have been working as a HO in their respective hospitals. The organisers will keep track of placements of all participants via social media applications as part of the course is still maintaining connections and informal training after the course has ended and as participants start the process of job application and working.

Ethical considerations

This study's approval for ethical clearance will be obtained from JETHIC COMMITTEE FOR RESEARCH INVOLVING HUMAN SUBJECT University Putra Malaysia ETHIC COMMITTEE FOR RESEARCH INVOLVING HUMAN SUBJECT (JKEUPM) ) and National Medical Research Register (NMRR); Medical Research and Ethics Committee (MREC) as the participants will be working in Ministry of Health facilities during the 1 month follow up. This study will also be registered in the National Institute of Health (NIH) as a trail registration.

Informed consent will be obtained from each study participant and they will be told the right not to respond to the questions they don't want to respond to or to withdraw from the study at any time. All data obtained will be kept confidentially and for research purposes only.

The benefits of the study includes assessing issues in relations to HO wellbeing and to assess what is needed in training a functional HO. The potential risk, discomforts and inconvenience is almost none. However, should the DASS score be suggestive of depression or anxiety, team members of the research team will refer the participant appropriately. Should participants choose to withdraw from study, they will be allowed to do so.

Data Analysis

The data will be analysed using IBM Social Package for Social Science (SPSS) version 24. A descriptive analysis of the demographic characteristics of the participants, clinical experience and baseline level of confidence, readiness and psychological wellbeing will be reported using means and standard deviations (SD) or median and inter-quartile range (IQR) for continuous variables (depending on the data distribution) and as frequencies and percentages for categorical data. An analysis to compare between participants who completed and withdrew from the study will be made using Chi-square or Exact test (for unbalanced data) for categorical variables and independent t-test for continuous data.

A repeated measures ANOVA will be conducted to determine the effectiveness of the intervention within the groups across the study periods (baseline, immediately after intervention and at 1 month after working). Controlling for baseline measures will be done to determine the change over time on the measured outcomes (level of confidence, readiness and psychological wellbeing). All analyses conducted are two-tailed with significant level set at p value <0.05.

Operational Definitions of terms

1. Medical Graduates/Participants - Those that have obtained a medical degree be it MD, MBBCh BAO, MBBS or the same level
2. Socio-demography - the components of description of a population

   1. Age - based on the year a person was born
   2. Sex- male or female
   3. Marital Status - single, married, separated or divorced
   4. Ethnicity - background of a person's race
   5. Religion - the religion based on identification card (I.C)
   6. Year of graduation - year they receive their certificates of qualification
   7. University- institution of higher learning they graduated from
   8. Confidence -a feeling of self-assurance arising from an appreciation of one's own abilities or qualities
   9. Readiness - the state of being fully prepared for something.
   10. Psychosocial well-being - the state of, affecting, or arising in the mind; related to the mental and emotional state of a person.

ELIGIBILITY:
Inclusion Criteria:

1. Participants that have registered to attend the Medicorp HO Preparatory Course

Exclusion Criteria:

1. Participants declared to have psychiatric illness
2. Participants who have not completed a medical degree (medical students)
3. Participants already working as a H

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aneesa Abdul Rashid, MBBCh BAO, Principal Investigator — UPM
Locations (1):
- FRIM, Kepong, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rashid AA, Shariff Ghazali S, Mohamad I, Mawardi M, Roslan D, Musa H. Quasi-experimental study on the effectiveness of a house officer preparatory course for medical graduates on self-perceived confidence and readiness: a study protocol. BMJ Open. 2019 Aug 10;9(8):e024488. doi: 10.1136/bmjopen-2018-024488. PMID 31401588

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants in Medicorp HO Preparatory Module: A total of 267 participants registered for the course and were invited to participate within the timeframe of this study period of recruitment. Only 239 returned their baseline questionnaires. At the time-point immediately after the intervention, 224 participants returned their completed questionnaires. At the subsequent follow up of the study, which was one-month post working as a HO, 101 answered the questionnaire.
Period: Overall Study
Arm/Group | Participants in Medicorp HO Preparatory Module
Started | 267
Completed | 101
Not Completed | 166

BASELINE CHARACTERISTICS:
Groups:
- Sociodemographic Factors of Participants: Data and results obtained from pre-intervention, post intervention and 1 month after work post intervention
Arm/Group | Sociodemographic Factors of Participants
Number analyzed (Participants) | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.66 (1.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186
  Male | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Malay | 189
  Chinese | 19
  Indian | 19
  Others | 12
Religion [Count of Participants; unit: Participants]
  Islam | 194
  Christian | 18
  Hindu | 16
  Buddha | 7
  Others | 4
Year of Graduation [Count of Participants; unit: Participants]
  2016 | 2
  2017 | 81
  2018 | 156
Place of Graduation [Count of Participants; unit: Participants]
  Local | 63
  Overseas | 176

OUTCOME MEASURES:

1. Primary Outcome: Change in Confidence Level
Description: This will be adapted from the IMU Student Competency Survey (Appendix 2) as there are no published studies on the confidence level of medical graduates before beginning HO-ship. The questionnaire comprises of 5 sections. The first 4 sections asses on generic skills, practical tasks, soft skills and their confidence as a whole, using a Likert scale assessment. Scoring is a mean score of 1-5 and the higher the score, the higher the confidence. The last section asks on the one daunting aspect of being a HO out of a list of 7 things, this section is descriptive.
Time Frame: pre intervention, immediately after intervention and 1 month after working as a House Officer ( an average of 6 months after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-intervention: The participants assessed before the preparatory course started.
- Post-intervention: The participant assessed after the preparatory course ended.
- Post 1 Month Working: The participant assessed after 1 month working.
Arm/Group | Pre-intervention | Post-intervention | Post 1 Month Working
Number analyzed (Participants) | 239 | 224 | 101
score on a scale | 2.18 (1.00) | 3.50 (0.75) | 3.79 (0.92)

2. Secondary Outcome: Change in Readiness Level
Description: This is also adapted from the IMU competency survey and is asked on a likert scale of 1 to 5 for their level of readiness. It is assessed after the confidence section. The higher the score, the higher the level of readiness
Time Frame: pre intervention, immediately post intervention (after 3 days of intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-intervention Level of Readiness: The participants assessed before the preparatory course started.
- Post Intervention Level of Readiness: The participants assessed after the preparatory course ended.
Arm/Group | Pre-intervention Level of Readiness | Post Intervention Level of Readiness
Number analyzed (Participants) | 239 | 224
score on a scale | 2.36 (1.03) | 3.46 (0.78)

3. Secondary Outcome: Change in Psychological Well Being - Depression
Description: This is using the Depression Anxiety Stress Scale (DASS): This questionnaire is used to asses Depression, Anxiety and Stress. It uses a likert scale. The scores indicate normal, mild, moderate, severe and extremely severe for each of the domains. The higher the scores, indicates the more severe the conditions.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia.
  Minimum score: 0 Maximum score: 42
  Normal: 0-9 Mild: 10-13 Moderate: 14-20 Severe: 21-27 Exteremely severe: 28+
Time Frame: pre intervention and 1 month after working as a House Officer ( an average of 6 months after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-intervention DASS-depression: The participant assessed before the preparatory course started via DASS questionnaire.
- Post 1 Month Working DASS-depression: The participants assessed after the preparatory course ended via DASS questionnaire.
Arm/Group | Pre-intervention DASS-depression | Post 1 Month Working DASS-depression
Number analyzed (Participants) | 239 | 101
score on a scale | 8.67 (7.93) | 7.80 (8.95)

4. Secondary Outcome: Change in Psychological Well Being - Anxiety
Description: This is using the Depression Anxiety Stress Scale (DASS): This questionnaire is used to asses Depression, Anxiety and Stress. It uses a likert scale. The scores indicate normal, mild, moderate, severe and extremely severe for each of the domains. The higher the scores, indicates the more severe the conditions.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect.
  Minimum score: 0 Maximum score: 48
  Normal: 0-7 Mild: 8-9 Moderate: 10-14 Severe: 15-19 Extremely severe: 20+
Time Frame: pre intervention and 1 month after working as a House Officer ( an average of 6 months after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-intervention DASS-anxiety: The participants assessed before the preparatory course via DASS questionnaire.
- Post 1 Month Working DASS-anxiety: The participants assessed 1 month after working via DASS questionnaire.
Arm/Group | Pre-intervention DASS-anxiety | Post 1 Month Working DASS-anxiety
Number analyzed (Participants) | 239 | 101
score on a scale | 9.75 (7.24) | 7.43 (9.54)

5. Secondary Outcome: Change in Psychological Well Being - Stress
Description: This is using the Depression Anxiety Stress Scale (DASS): This questionnaire is used to asses Depression, Anxiety and Stress. It uses a likert scale. The scores indicate normal, mild, moderate, severe and extremely severe for each of the domains. The higher the scores, indicates the more severe the conditions.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content The stress scale is sensitive to levels of chronic non-specific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.
  Minimum score: 0 Maximum score: 48
  Normal: 0-14 Mild: 15-18 Moderate: 19-25 Severe: 26-33 Extremely severe: 34+
Time Frame: pre intervention and 1 month after working as a House Officer ( an average of 6 months after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-intervention DASS-stress: The participants assessed before the preparatory course via DASS questionnaire.
- Post 1 Month Working DASS-stress: The participants assessed 1 month after working via DASS questionnaire.
Arm/Group | Pre-intervention DASS-stress | Post 1 Month Working DASS-stress
Number analyzed (Participants) | 239 | 101
score on a scale | 11.78 (8.05) | 8.58 (10.33)

ADVERSE EVENTS:
Time Frame: 1 year
Description: This is an education module, hence, there should be no adverse events. However, in the module there were needle used in practical session. Therefore, needle prick injury can be one of the adverse events that we can include in the study.
  The adverse event is somehow monitored but not observed.
Groups:
- Participants in Medicorp HO Preparatory Module: Pre-intervention: The participants screened based on the exclusion and inclusion criteria leaving the number of 239 participants after registration.
  Post-intervention: Drop outs mainly due to failure in submitting the complete post-intervention questionnaires before they headed home.
  Post 1 month after work: Major drop outs purely as a result of unavailability to answer and time constraint due to the hectic schedule of a houseman.
Arm/Group | Participants in Medicorp HO Preparatory Module
All-Cause Mortality (participants affected / at risk) | 0/239
Serious Adverse Events (participants affected / at risk) | 0/239
Other Adverse Events (participants affected / at risk) | 0/239

LIMITATIONS AND CAVEATS:
Poor responses from the participants during follow-ups. Many of the participants are also lost to follow up made the number of drop outs bigger.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT03510195/Prot_SAP_000.pdf